CLINICAL TRIAL: NCT04944602
Title: A Multicenter Randomized, Double-blind, Parallel, Positive-controlled Phase III Clinical Trial to Evaluate the Therapeutic Equivalence of SYN008 Versus Xolair® in the Treatment of Patients With Refractory Chronic Spontaneous Urticaria
Brief Title: Study to Evaluate the Therapeutic Equivalence of SYN008 Versus Xolair® in the Treatment of Patients With Refractory Chronic Spontaneous Urticaria
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC Baike (Shandong) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYSA1903-CSP-002
Record Dates: First submitted 2021-06-09; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — Omalizumab; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYN008 (Experimental): patients received a dose of SYN008 300 mg which consisted of two injections of omalizumab 150 mg vials every 4 weeks (Day 1, Week 4 and Week 8)
  Interventions: Biological: SYN008
- Omalizumab (Active Comparator): patients received a dose of omalizumab 300 mg which consisted of two injections of omalizumab 150 mg vials every 4 weeks (Day 1, Week 4 and Week 8)
  Interventions: Biological: Omalizumab for injection

INTERVENTIONS:
Biological: SYN008 — injection of 300 mg
  Arms: SYN008
Biological: Omalizumab for injection — injection of 300 mg
  Arms: Omalizumab

SUMMARY:
• This study is a multicenter, randomized, double-blind, parallel-group, positive-controlled phase III study to evaluate the therapeutic equivalence of SYN008 versus omalizumab for injection (Xolair®) in the treatment of CSU patients who remain symptomatic despite antihistamine treatment.

DETAILED DESCRIPTION:
A total of approximately 340 patients with H1 antihistamines (H1AH) refractory CSU will be randomized into two treatments arms (SYN008 300 mg s.c., and omalizumab 300 mg s.c.) at a 1:1 ratio. Both SYN008 and omalizumab will be injected every 4 weeks as an add-on therapy on top of H1AH treatment.

The study will consist of three distinct epochs over 27 weeks, as follows:

* Screening epoch: Day -21 to Day -1
* Randomized-treatment epoch: Day 1 to Week 12
* Post-treatment follow-up epoch: Week 1

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CSU refractory to H1AH at the time of randomization, as defined by all of the following:

   * CSU diagnosis for ≥ 6 months;
   * The presence of itch and hives for ≥ 6 consecutive weeks within one year prior to randomization despite use of H1AH treatment during this time period;
   * UAS7 score (range 0-42) ≥ 16 and itch component of UAS7 (range 0-21) ≥ 8 during 7 days prior to randomization (Day 1);
   * In-clinic UAS ≥ 4 on at least one of the screening visit days;
   * Patients must have been on an approved dose of an H1AH for CSU for at least the 3 consecutive days immediately prior to the screening visit and must have documented current use on the day of the initial screening visit.
2. Voluntarily sign the informed consent form. Willing and able to complete a daily symptom diary for the duration of the study, and comply with the protocol requirements.
3. Patients must not have had any missing diary entries in the 7 days prior to randomization.
4. Both male and female patients must agree to practice contraception from the signing of informed consent to 6 months after the last dose of study drugs.

Exclusion Criteria:

1. Previous treatment with omalizumab within one year prior to signing the informed consent.
2. Hypersensitivity to omalizumab, study drug excipients or other biosimilars, or have a history of severe drug allergy or anaphylactic shock.
3. Clearly defined underlying etiology for chronic urticarias other than CSU. This includes but is not limited to:

   1. dermatographism (factitious urticaria);
   2. cold, heat, solar, delayed pressure, aquagenic, cholinergic or contact urticarias;
   3. Any of the following diseases, which may have symptoms of urticaria and/or angioedema: urticarial vasculitis, urticaria pigmentosa, erythema multiforme, mastocytosis, hereditary or acquired angioedema, lymphoma, leukemia, etc.
4. Patients with a stool examination positive for ova or parasites at screening. {Stool ova and parasite evaluation will only be conducted in patients with BOTH risk factors for parasitic disease (living in an endemic area, and/or chronic gastrointestinal (GI) symptoms and chronic immunosuppression, travel within the last 6 months to an endemic area) AND an absolute eosinophil count more than twice the upper limit of normal.}
5. Suffer from other chronic pruritic dermatosis that may confound the results: atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, senile pruritus, etc.
6. CSU patients who had difficulty breathing episodes due to angioedema in the past six months.
7. Active infections requiring treatment at screening, include but not limited to pulmonary infection and tuberculosis.
8. Patients with platelet count ≤100*109/L at screening.
9. A history of malignancy of any organ or system within 5 years prior to screening, regardless of local recurrence or metastasis {except for basal cell carcinoma, actinic keratosis, or Bowen's disease (squamous cell carcinoma in situ) that have been treated and have not recurred in the past 12 weeks; Cervical carcinoma in situ or non-invasive malignant colonic polyps that have been resected and have not recurred within the last 5 years}
10. Presence of clinically significant unstable diseases:

    * High risk of severe ventricular arrhythmias, such as significant left ventricular dysfunction, NYHA class III / IV;
    * Myocardial infarction occurred within 6 months before screening. History of unstable angina, acute coronary syndrome or other high-risk coronary heart disease;
    * Poorly controlled hypertension [Hypertension diagnosis of grade II or III, high risk, and systolic blood pressure (SBP) ≥ 160 mmHg or diastolic blood pressure (DBP) ≥ 100 mmHg while taking one or two antihypertensive drugs].
11. Presence of clinically significant cardiovascular, neurological, psychiatric, metabolic, hepatic, or other pathological conditions that could interfere with the interpretation of the study results and or compromise the safety of the patients, e.g.:

    * Abnormal liver function [AST or ALT ≥ 1.5 x ULN, or total bilirubin ≥ 1.5 x ULN]; abnormal renal function [elevated serum creatinine > 1.5 x ULN];
    * HBsAg positive and HBV DNA quantitative value exceeds the upper limit of the normal value range of each research site, or positive in any one of the tests of hepatitis C virus antibody, HIV antibody and Treponema pallidum antibody;
    * ECG abnormalities of clinical significance, e.g., clinically significant II-III degree atrioventricular (AV) block without a pacemaker, QTc interval≥480 ms, or sustained tachycardia requiring treatment.
12. History of alcohol or drug abuse, within the last 6 months prior to screening.
13. Currently participating in other clinical trials, or have received any experimental intervention within 3 months prior to signing the informed consent.
14. Pregnant or nursing (lactating) women.
15. Currently taking or plan to take medications prohibited by the protocol at screening.
16. Other conditions deemed by investigator as unsuitable for this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
The change from baseline in the Weekly Itch Severity Score (ISS7) at week 12 | week 12
  The severity of the itch was recorded by the patient twice daily in their Diary, on a scale of 0 (none) to 3 (intense/severe). Baseline ISS7 was calculated 7 days prior to the first treatment date. A weekly score (ISS7) was derived by adding up the average daily scores of the seven days preceding the visit. The possible range of the weekly score was therefore 0 to 21, where 0 is the best score and 21 is the worst score. The complete itch response was defined as ISS7 = 0.
  Itch (Pruritus) Severity Score Scale:
  0 = None
  1. = Mild (minimal awareness, easily tolerated)
  2. = Moderate (definite awareness, bothersome but tolerable)
  3. = Severe (difficult to tolerate)

SECONDARY OUTCOMES:
The change from baseline in Urticaria Activity Score Over 7 Days (UAS7) at week 12 | week 12
  UAS7 is the sum of the NHS7 and the ISS7 scores. The possible range of the weekly UAS7 score is 0 to 42. A higher urticaria activity score indicates more severe symptoms. A negative change score from baseline indicates improvement.
The change from baseline in Weekly Number of Hives Score (NHS7) at week 12 | week 12
  Hives Severity Score (HSS), defined by number of hives, were recorded by the patient once daily in their Diary, on a scale of 0 (none) to 3 (intense/severe). A weekly number of hives score (NHS7) was derived by adding up the average daily scores of the seven days preceding the visit. The possible range of the weekly score was therefore 0 to 21. The complete hives response was defined as NHS7 = 0.
  Hives Severity Score scale:
  0 = None
  1. = Mild
  2. = Moderate
  3. = Severe
Percentage of patients with UAS7≤6 | week 12
  UAS7 is the sum of the NHS7 and the ISS7 scores. The possible range of the weekly UAS7 score is 0 to 42. A higher urticaria activity score indicates more severe symptoms. A negative change score from baseline indicates improvement. Week 12 responders were defined as patients who achieved an absolute UAS7 ≤ 6 at Week 12. A patient with missing data at Week 12 was imputed as a responder if the patient was a responder at Week 10 and Week 11, otherwise as a non-responder.
Correlation analysis between baseline changes of ISS7/UAS7 and baseline IgE level | week 12
  The weekly itch severity score is the sum of the daily itch severity scores over 7 days. UAS7 is the sum of the NHS7 and the ISS7 scores.A negative change score from baseline indicates improvement. CSU patients' baseline IgE level correlates with the improvement to a certain extent.
Time to ISS7 minimal important differences (MID) response | week 12
  The weekly itch severity score is the sum of the daily itch severity scores over 7 days and ranges from 0 to 21. The daily itch severity score is the average of the morning and evening scores on a scale of 0 (none) to 3 (severe). The Baseline weekly itch severity score is the sum of the daily itch severity scores over the 7 days prior to the first treatment. A higher itch severity score indicates more severe itching. A negative change score indicates improvement.
  The MID response for weekly itch severity score was defined as a reduction from baseline in weekly itch severity score of 5 points or more. The time to weekly itch severity score MID response was defined as the time (in weeks) from Day 1 to the study week when weekly itch severity score MID response was first achieved.
Percentage of patients with ISS7 MID response | week 12
  The MID response for weekly itch severity score was defined as a reduction from baseline in weekly itch severity score of 5 points or more. This outcome measure shows the percentage of participants classified as MID Responders at Week 12, meaning their weekly itch severity scores at Week 12 were at least 5 points lower than at Baseline.
Change from baseline in Overall Dermatology Life Quality Index (DLQI) score | week 12
  Dermatology life quality index (DLQI) is a 10-item dermatology- specific health-related quality of life measure. Patients rated their dermatology symptoms as well as the impact of their skin condition on various aspects of their lives. An overall score was calculated as well as separate scores for the following domains: symptoms and feelings, daily activities, leisure, work and school, personal relationships, treatment. Each domain had 4 response categories ranging from 0 (not at all) to 3 (very much). "Not relevant" is a valid score also and is scored as 0. The DLQI total score is a sum of all 10 responses. Scores range from 0 to 30 with higher scores indicating greater health-related quality of life impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Ruo-Yu Li, Principal Investigator — Peking University First Hospital

IPD SHARING:
Plan to Share IPD: No